CLINICAL TRIAL: NCT01621191
Title: An Open Label Extension Study of Phase 3 Trial of Duloxetine in Patients With Fibromyalgia
Brief Title: An Extension Study of Duloxetine in Fibromyalgia (Extension of F1J-JE-HMGZ, NCT01552057)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14614; F1J-JE-HMHB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 60 mg Duloxetine (Experimental): Duloxetine 20 milligrams (mg) taken orally once every day for 1 week, followed by 40 mg taken orally once every day for 1 week, and then 60 mg taken orally once every day for 48 weeks
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Administered Orally
  Other Names: LY248686; Cymbalta; Ariclaim; Xeristar; Yentreve

SUMMARY:
The purpose of the study is to assess the safety and efficacy of duloxetine in participants with fibromyalgia at long-term use.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the 15-week treatment in the preceding study HMGZ
* Participants who wish continuous treatment with duloxetine after the preceding study
* Participants are able to give their own written consent

Exclusion Criteria:

* Participants with serious cardiovascular, hepatic, renal, respiratory, or hematological disease, or clinically significant laboratory or electrocardiogram abnormality which indicate a serious medical problem or require significant intervention in the judgment of the investigators
* Participants with alanine aminotransferase/aspartate aminotransferase of not less than 100 International Units/Liter (IU/L) or total bilirubin of not less than 1.6 milligrams/deciliter (mg/dL) at Week 0 (Visit 8 of the preceding study)
* Participants with serum creatinine level of not less than 2.0 mg/dL, participant who has undergone kidney transplantation or hemodialysis at Week 0 (Visit 8 of the preceding study)
* Participants with pain difficult to discriminate from pain associated with fibromyalgia or disease which disturbs the assessment
* Participants with thyroidal dysfunction, excluding those assessed by the investigator that the disorder is controlled as appropriate by three-month or longer drug therapy
* Participants with present or past history of rheumatoid arthritis, inflammatory arthritis, infectious arthritis, or auto immune disease rather than thyroid deficiency
* Participants with uncontrolled angle closure glaucoma
* Participants who received monoamine oxidase (MAO) inhibitors within 14 days before Week 0 (Visit 8 of the preceding study) or need to receive a MAO inhibitor within 5 days after study discontinuation
* Participants who have experienced suicidal ideation or suicide attempt during the preceding study
* Participants answering "yes" to any of the questions about active suicidal ideation/intent/behaviors occurring in the preceding study (Columbia Suicide Severity Rating Scale, Suicide Ideation section - Questions 4 and 5; Suicidal Behavior section)
* Female participants who are pregnant, lactating, or who want to get pregnant during the study period. Male participants who want his partner to get pregnant
* Females of child-bearing potential who cannot agree to utilize medically acceptable and reliable means of birth control during the study and for 1 month following the last dose of the study
* Participants assessed ineligible by the investigator (sub-investigator) for other reasons

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the 15-week treatment in the preceding study F1J-JE-HMGZ (HMGZ) (NCT01552057) were enrolled in this study.
Pre-assignment Details: Enrolled participants who completed the 50-week treatment period were considered to have completed the study. After study completion or early discontinuation, participants completed a 2-week taper and were observed 1 week post-treatment for safety.
Groups:
- Duloxetine 60 mg: Treatment Period: Up to a 60-milligram (mg) dose of duloxetine was administered orally once daily for 50 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule), Week 2: 40-mg dose of duloxetine (two 20-mg capsules), and Weeks 3 through 50: 60-mg dose of duloxetine (three 20-mg capsules).
  During the 2-week taper, the daily dosage was gradually reduced. For the first week: 40-mg dose of duloxetine (two 20-mg capsules) administered orally once daily. For the second week: 20-mg dose of duloxetine (one 20-mg capsule) administered orally once daily.
Period: Overall Study
Arm/Group | Duloxetine 60 mg
Started | 149
Received at Least 1 Dose of Study Drug | 149
Had at Least 1 Post-Baseline Observation | 148
Completed | 124
Not Completed | 25
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 8
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 1
Not completed — Site Removed From Study | 1

BASELINE CHARACTERISTICS:
Population: Enrolled participants who received at least 1 dose of study drug and had at least 1 post-baseline observation.
Groups:
- Duloxetine 60 mg: Treatment Period: Up to a 60-mg dose of duloxetine was administered orally once daily for 50 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule), Week 2: 40-mg dose of duloxetine (two 20-mg capsules), and Weeks 3 through 50: 60-mg dose of duloxetine (three 20-mg capsules).
  During the 2-week taper, the daily dosage was gradually reduced. For the first week: 40-mg dose of duloxetine (two 20-mg capsules) administered orally once daily. For the second week: 20-mg dose of duloxetine (one 20-mg capsule) administered orally once daily.
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 148
Region of Enrollment [Number; unit: participants]
  Japan | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 53 weeks
Population: Enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 149
participants | 138

2. Secondary Outcome: Patient Global Impression-Improvement (PGI-I) at Endpoint
Description: PGI-I measures the participant's perception of improvement at the time of assessment compared with the start of treatment. Scores ranged from 1 (very much better) to 7 (very much worse).
Time Frame: 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 PGI-I assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine 60 mg: Treatment Period: Up to a 60-mg dose of duloxetine was administered orally once daily for 50 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule), Week 2: 40-mg dose of duloxetine (two 20-mg capsules), and Weeks 3 through 50: 60-mg dose of duloxetine (three 20-mg capsules).
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale | 2.48 (1.31)

3. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) at Endpoint
Description: CGI-I measures the clinician's perception of participant improvement at the time of assessment (compared with the start of treatment). Scores ranged from 1 (very much better) to 7 (very much worse).
Time Frame: 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 CGI-I assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale | 2.34 (1.08)

4. Secondary Outcome: Change From Baseline to 50-Week Endpoint in Fibromyalgia Impact Questionnaire (FIQ)
Description: FIQ is a 20-item, self-administered questionnaire using Likert-type scales to measure participant outcomes over the past week. Items 1 through 11 measured physical functioning on 4-point scales. Items 12 and 13 measured the number of days a participant felt well and days a participant was unable to work due to fibromyalgia symptoms, respectively. Items 14 through 20 were 11-point scales on which a participant rated work difficulty, pain, fatigue, morning tiredness, stiffness, anxiety, and depression, respectively. If a participant did not do all the tasks listed, those items were deleted from scoring. Algorithms were used to determine total FIQ scores which ranged from 0 to 100; higher scores indicated a more negative impact.
Time Frame: Baseline, 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 FIQ assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale | -6.00 (15.12)

5. Secondary Outcome: Change From Baseline to 50-Week Endpoint in Brief Pain Inventory-Severity (BPI-S) and Brief Pain Inventory-Interference (BPI-I) Scores on the BPI-Modified Short Form
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function, respectively. Severity scores ranged from 0 (no pain) to 10 (severe pain) for each question assessing average pain, worst pain, least pain, and pain right now. Interference scores ranged from 0 (does not interfere) to 10 (completely interferes) for each question assessing interference of pain in past 24 hours with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference was the average of non-missing scores of individual interference items.
Time Frame: Baseline, 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 BPI-S or BPI-W assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale
  Average Pain | -1.31 (1.70)
  Worst Pain | -1.53 (1.87)
  Least Pain | -1.26 (1.82)
  Pain Right Now | -1.47 (2.03)
  Interference With General Activity | -0.72 (2.04)
  Interference With Mood | -0.82 (1.82)
  Interference With Walking Ability | -0.73 (2.04)
  Interference With Normal Work | -0.66 (2.01)
  Interference With Relations With Other People | -0.38 (1.95)
  Interference With Sleep | -1.00 (2.26)
  Interference With Enjoyment of Life | -0.68 (2.00)
  Average Interference | -0.71 (1.65)

6. Secondary Outcome: Change From Baseline to 50-Week Endpoint in 36-Item Short-Form (SF-36) Health Survey Domain Scores
Description: The SF-36 Health Survey is a generic, health-related survey assessing the participant's quality of life on 8 domains: physical functioning, daily functioning (physical), bodily pain, general health, vitality, social functioning, daily functioning (emotional), and mental health. Each domain was scored by summing individual items pertaining to that domain and transforming scores into a 0 to 100 scale, with higher scores indicating better health status or functioning.
Time Frame: Baseline, 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 SF-36 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale
  Physical Functioning | 4.26 (14.54)
  Role-Physical | 4.02 (17.05)
  Bodily Pain | 6.89 (14.89)
  General Health | 4.14 (11.88)
  Vitality | 0.16 (18.13)
  Social Functioning | 3.26 (21.47)
  Role-Emotional | 3.55 (18.83)
  Mental Health | 2.13 (14.00)

7. Secondary Outcome: Change From Baseline to 50-Week Endpoint in Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item self-administered questionnaire designed to assess the characteristics of depression. Each item was scored on a 4-point scale ranging from 0 (not present) to 3 (present in the extreme) and was summed to give a total BDI-II score. A total BDI-II score of 0 through 13 was considered minimal, 14 through 19 was mild, 20 through 28 was moderate, and 29 through 63 was severe depression symptoms.
Time Frame: Baseline, 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 BDI-II assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale | -0.94 (5.22)

8. Secondary Outcome: Change From Baseline to 50-Week Endpoint in Widespread Pain Index (WPI) and Symptom Severity (SS) in American College of Rheumatology (ACR) Fibromyalgia Diagnostic Criteria 2010
Description: WPI: Participant-reported areas (out of 19 points on the body) in which the participant had pain in the past week. WPI scores ranged from 0 (no areas) to 19 (all areas). SS: The sum of severity scores for fatigue, waking unrefreshed, and cognitive symptoms [each rated from 0 (no problem) to 3 (severe; life-disturbing problems)] plus the severity of somatic symptoms in general [rated from 0 (no symptoms) to 3 (a great deal of symptoms)]. The total SS score ranged from 0 and 12.
Time Frame: Baseline, 50 weeks
Population: Enrolled participants who received at least 1 dose of study drug and had a Week 50 WPI or SS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 60 mg
Number analyzed (Participants) | 115
units on a scale
  WPI | -1.46 (3.74)
  SS | -0.37 (1.27)

ADVERSE EVENTS:
Time Frame: Baseline through 53 weeks
Groups:
- 60 mg Duloxetine: Treatment Period: Up to a 60-mg dose of duloxetine was administered orally once daily for 50 weeks. During the first 2 weeks of treatment, participants gradually increased their dosage. Week 1: 20-mg dose of duloxetine (one 20-mg capsule), Week 2: 40-mg dose of duloxetine (two 20-mg capsules), and Weeks 3 through 50: 60-mg dose of duloxetine (three 20-mg capsules).
  During the 2-week taper, the daily dosage was gradually reduced. For the first week: 40-mg dose of duloxetine (two 20-mg capsules) administered orally once daily. For the second week: 20-mg dose of duloxetine (one 20-mg capsule) administered orally once daily.
Arm/Group | 60 mg Duloxetine
Serious Adverse Events (participants affected / at risk) | 8/149
Other Adverse Events (participants affected / at risk) | 138/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 60 mg Duloxetine (N=149)
Retinal detachment (Eye disorders) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1)
Self injurious behaviour (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 60 mg Duloxetine (N=149)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Bundle branch block left (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4)
Prinzmetal angina (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 9 (9)
Blepharitis allergic (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 2 (2)
Corneal degeneration (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Scleral haemorrhage (Eye disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 5 (7)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9)
Constipation (Gastrointestinal disorders) | 27 (31)
Dental caries (Gastrointestinal disorders) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (5)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 3 (3)
Large intestine polyp (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (24)
Periodontal disease (Gastrointestinal disorders) | 3 (3)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Asthenia (General disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 5 (5)
Fatigue (General disorders) | 2 (2)
Feeling abnormal (General disorders) | 4 (4)
Local swelling (General disorders) | 2 (2)
Malaise (General disorders) | 8 (8)
Oedema (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Submandibular mass (General disorders) | 1 (1)
Thirst (General disorders) | 11 (11)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 9 (10)
Body tinea (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4)
Cystitis (Infections and infestations) | 6 (6)
Gastroenteritis (Infections and infestations) | 3 (4)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Gingivitis (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 2 (3)
Infected dermal cyst (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 6 (6)
Nasopharyngitis (Infections and infestations) | 58 (102)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 5 (6)
Paronychia (Infections and infestations) | 4 (5)
Periodontitis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pertussis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 5 (5)
Pulpitis dental (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3)
Subcutaneous abscess (Infections and infestations) | 1 (2)
Tinea infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (7)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 6 (8)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 5 (6)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 2 (2)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (6)
Blood cholesterol increased (Investigations) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 4 (5)
Blood uric acid increased (Investigations) | 2 (2)
Eosinophil count increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 7 (8)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 2 (2)
Weight increased (Investigations) | 14 (14)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myofascitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Autonomic neuropathy (Nervous system disorders) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (10)
Dysgeusia (Nervous system disorders) | 2 (2)
Head discomfort (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (9)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1)
Parosmia (Nervous system disorders) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1)
Radial nerve palsy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 34 (34)
Visual field defect (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9)
Nightmare (Psychiatric disorders) | 3 (3)
Somatoform disorder gastrointestinal (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/122 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1/122 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 7 (7)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days